CLINICAL TRIAL: NCT06805825
Title: A Phase 1 Dose Escalation and Expansion Study of the c-Kit Specific Antibody-Drug Conjugate NN3201 in Subjects With Advanced and/or Metastatic Solid Tumors Known to Express c-Kit
Brief Title: A Study of the c-Kit Specific Antibody-Drug Conjugate NN3201 for Advanced and/or Metastatic Solid Tumors Known to Express c-Kit
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novelty Nobility, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NN3201-ST100
Record Dates: First submitted 2025-01-08; First posted 2025-02-03 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Gastrointestinal Stromal Tumors; Small-cell Lung Cancer; Adenoid Cystic Carcinoma; Uveal Melanoma; Neuroendocrine Tumors; Chromophobe Renal Cell Carcinoma; Clear Cell Renal Cell Carcinoma
Keywords: GIST; SCLC; ACC; NET; ChRCC; ccRCC; Novelty Nobility; cKit; c-kit; Gastrointestinal Stromal Tumors; Small-cell Lung Cancer; Adenoid Cystic Carcinoma; Uveal Melanoma; Neuroendicrine Tumors; Chromophobe Renal Cell Carcinoma; Clear Cell Renal Cell Carcinoma; advanced GIST; advanced SCLC; advanced ACC; advanced NET; advanced ChRCC; advanced ccRCC
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Small Cell Lung Carcinoma; Carcinoma, Adenoid Cystic; Uveal Melanoma; Neuroendocrine Tumors; Carcinoma, Renal Cell; Piebaldism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part A (Experimental): NN3201 administered intravenously every three weeks, the dosage to be determined by ascending dose cohort assignment. Part A will enroll patients that have GIST or Other c-Kit tumor disease types. This is an open-label multiple ascending dose study.
  Interventions: Drug: NN3201
- Part B, Cohort 1 (GIST) (Experimental): NN3201 administered intravenously every three weeks, expanding one or two doses in GIST disease type. This is an open-label multiple dose expansion study.
  Interventions: Drug: NN3201
- Part B, Cohort 2 (SCLC) (Experimental): NN3201 administered intravenously every three weeks, expanding one or two doses in SCLC disease type. This is an open-label multiple dose expansion study.
  Interventions: Drug: NN3201
- Part B, Cohort 3 (other c-Kit tumors) (Experimental): NN3201 administered intravenously every three weeks, expanding one or two doses in Other c-Kit tumor disease type. This is an open-label multiple dose expansion study.
  Interventions: Drug: NN3201

INTERVENTIONS:
Drug: NN3201 — A c-Kit targeting fully human monoclonal antibody-drug conjugate with MMAE administered intravenously.

SUMMARY:
This open-label clinical trial will evaluate the safety and tolerability of NN3201 in subjects with advanced and/or metastatic solid tumors known to express c-Kit.

DETAILED DESCRIPTION:
The drug being tested in this study is called NN3201, a c-Kit targeting fully human monoclonal antibody-drug conjugate with MMAE, administered by IV. The study will be conducted in two parts, a dose escalation phase (Part A) followed by an expansion phase (Part B).

The patient population for the dose escalation phase (Part A) of the study will include patients with advanced and/or metastatic c-Kit-associated solid tumors including gastrointestinal stromal tumor (GIST), adenoid cystic carcinoma (ACC), uveal melanoma, neuroendocrine tumors (NET), and chromophobe and clear cell renal cell carcinomas (ChRCC and ccRCC). For Part A patients must have received treatment with imatinimb for GIST or be progressive/refractory, ineligible, or intolerant to available standard therapy (or subject declines standard therapy) for cKit-associated solid tumors (ACC, uveal melanoma, NET, ChRCC, or ccRCC). The primary objective of the dose escalation phase (Part A) is to determine the safety profile of NN3201 administered by IV, including the incidence and severity of adverse events (AEs), serious adverse events (SAEs), and dose-limited toxicities (DLTs) as well as the incidence of abnormal laboratory findings and abnormal vital signs. Part A will help determine the maximum tolerated dose (MTD) and/or the recommended dose(s) (RDEs) for the expansion phase (Part B).

Once a recommended dose has been determined in the escalation phase (Part A), the expansion phase (Part B) will assess the safety and efficacy of NN3201 when administered at 2 RDE dose levels to subjects in two indication-specific (GIST and SCLC) expansion cohorts and one basket cohort for c-Kit positive solid tumors (excluding GIST and SCLC). All cohorts in Part B will utilize the same eligibility criteria as in Part A.

Cohort B1 - GIST: up to 10 subjects with GIST will be enrolled at the MTD level (RDE1) and efficacy and safety as well as any available PK and PD data will be evaluated.

Cohort B2 - SCLC: up to 10 SCLC will be enrolled at 1 dose level below MTD (MTD-1/RDE2) and efficacy and safety as well as any available PK and PD data will be evaluated. The Scientific Review Committee (SRC) may decide to enroll and additional 10 subjects in SCLC subjects.

Cohort B3 - c-Kit-associated solid tumors: in this basket cohort, up to 10 subjects with any c-Kit-associated solid tumor (including ACC, uveal melanoma, NET, ChRCC, and ccRCC and excluding GIST and SCLC) will be enrolled.

The safety and tolerability of NN3201 administered intravenously (IV) at up to two RDEs in subjects with advanced and/or metastatic solid tumors is the primary objective for Part B.

ELIGIBILITY:
Key Inclusion Criteria:

Subjects must meet the following criteria to be eligible for enrollment into the study:

1. Histologically or cytologically confirmed locally advanced, metastatic, and/or unresectable GIST, SCLC, ACC, uveal melanoma, NET ChRCC or ccRCC.
2. Subjects must have received the following treatment:

   Part A (Dose Escalation):

   i. Treatment with imatinib for GIST (at least one line of therapy with imatinib)

   or

   ii. Progressive/refractory, ineligible, or intolerant to available standard therapy (or subject declines standard therapy) for c-Kit-associated solid tumors (ACC, uveal melanoma, NET ChRCC or ccRCC)

   Part B (Dose Expansion):

   i. Treatment with imatinib for GIST (at least one line of therapy with imatinib) or

   ii. Progressive/refractory, ineligible, or intolerant to available standard therapy (or subject declines standard therapy) for Extensive stage SCLC or

   iii. Progressive/refractory, ineligible, or intolerant to available standard therapy (or subject declines standard therapy) for c-Kit-associated solid tumors (ACC, uveal melanoma, NET or ChRCC or ccRCC).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy ≥ 3 months before starting NN3201 in the opinion of the Investigator.
5. Age ≥ 18 years.
6. Laboratory values demonstrating adequately functioning kidney, liver and bone marrow (hematology).
7. Adequate heart function as measured by ECHO/MUGA scan.
8. Time between prior anticancer therapy including investigational agents and first dose of NN3201 as below:

   1. Cytotoxic chemotherapy - At least 21 days
   2. Non-cytotoxic chemotherapy (e.g., small molecule inhibitor) - At least 14 days
   3. Nitrosoureas - At least 6 weeks
   4. Monoclonal antibody(ies) - At least 28 days
   5. Radiotherapy - At least 14 days from local site radiation therapy
9. Negative Serum/urine pregnancy test (for subjects of childbearing potential)
10. All subjects of childbearing potential must agree to use contraception throughout the study and for additional 120 days after the last dose of assigned treatment. Subjects must refrain from donating sperm during the same period or Subjects who do not have childbearing potential are confirmed post-menopausal or sterile.
11. Voluntary agreement to provide written informed consent and have willingness and ability to comply with all aspects of the protocol.

Key Exclusion Criteria:

1. Has received prior therapy with a c-Kit agent (except GIST subjects).
2. Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms.
3. A condition requiring systemic treatment with corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to administration of study drugs (inhaled corticosteroids are allowed).
4. Any prior treatment-related (i.e., chemotherapy, immunotherapy, radiotherapy) clinically significant toxicities that have not resolved to Grade ≤ 1 or prior treatment-related toxicities that are clinically unstable and clinically significant at Study Entry, Day -2 to Cycle 1 Day 1.
5. Major surgery within 30 days before the first dose of study drug treatment in Cycle 1 on Day 1 (port placement for venous access is not considered major surgery).
6. Significant cardiovascular impairment.
7. Significant screening electrocardiogram (ECG) abnormalities.
8. Known active and clinically significant bacterial, fungal, or viral infection.
9. Uncontrolled hypertension defined as systolic blood pressure ≥ 160mmHg and/or diastolic blood pressure ≥ 100mmHg, despite optimal medical management.
10. Venous thrombosis or pulmonary embolism within the last 3 months prior to the screening.
11. Ongoing or active infection requiring intravenous treatment with anti-infective therapy or systemic therapy and/or any identified active COVID-19 infection.
12. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the subject's participation in this study.
13. People who are pregnant or breastfeeding.

Other inclusion and exclusion criteria must also be met to be eligible to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Dose-limiting Toxicities: | 3 weeks
  A DLT is defined as an AE that meets at least one of the criteria listed in protocol, according to National Cancer Institute (NCI) common terminology criteria for AE (CTCAE) version 5.0 and is considered by the investigator to be clinically relevant and attributed to the study treatment during the first 21 days after the first dose of study treatment.
Incidence of Adverse Events: | 1 year
  Number of subjects with adverse events (AEs) according to severity, seriousness, and relationship to study drug

SECONDARY OUTCOMES:
Choose which dose(s) will be used in the expansion cohorts | 1 year
  Assessing which dose(s) have anti-tumor benefit and an acceptable incidence of adverse events that allow for continued enrollment
Pharmacokinetics (PK) of NN3201 | 3 years
  Pharmacokinetics (PK) of NGM120 by measuring serum concentration of NGM120 at specified timepoints
Assessment of anti-tumor activity | 3 years
  Assessment of anti-tumor activity by RECIST 1.1
Choose which dose(s) may be used in a future study | 3 years
  Assessing which dose(s) have anti-tumor benefit and an acceptable incidence of adverse events that may be used in a future study.

OTHER OUTCOMES:
Immunogenicity against NN3201 | 3 years
  Immunogenicity against NN3201 by measuring percentage of subjects to develop antidrug antibodies and neutralizing antibodies
Correlation Between Pharmacokinetic (PK) and Pharmacodynamic (PD) Variables, Safety, and Efficacy | 3 yeas
  Evaluation of the correlation between PK parameters (e.g., Cmax, AUC) and PD effects (e.g., changes in target biomarkers), and their relationship to safety outcomes (e.g., incidence of adverse events) and efficacy outcomes (e.g., objective response rate and progression-free survival).
Changes in Biomarker Levels in Response to Treatment | At baseline and specified intervals over 3 years.
  Investigation of changes in specific biomarkers (e.g., soluble c-Kit) during treatment to assess their relationship to treatment response.
Correlation Between Baseline Biomarker Levels and Clinical Response/Toxicity | 3 years
  Assessment of the relationship between baseline levels of specific biomarkers (e.g., soluble c-Kit, tumor c-Kit expression) and clinical outcomes, including response to treatment and incidence of toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Sharma, MD, Principal Investigator — Novelty Nobility
Locations (5):
- United States (5):
  - University of Michigan Hospitals, Ann Arbor, Michigan
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No